CLINICAL TRIAL: NCT06031974
Title: Dietary Intervention to Stop Coronary Atherosclerosis in Computed Tomography: Long-Term Follow-Up
Acronym: DISCO-CT2
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: 2.25/III/23
Record Dates: First submitted 2023-04-25; First posted 2023-09-11 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease; Diet, Healthy; Lifestyle Risk Reduction
MeSH Terms: conditions — Coronary Artery Disease; Risk Reduction Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DISCO Intervention: Patients included to the DISCO-CT study and randomized to the experimental arm, ie. subjected to optimal medical treatment in accordance with European Society of Cardiology recommendations + DASH diet (Dietary Approaches to StopHypertension) and strict monitoring of eating and lifestyle behaviors
  n=46
  Interventions: Behavioral: DISCO Intervention
- Control: Patients included to the DISCO-CT study and randomized to the control arm, ie. subjected to optimal medical treatment in accordance with European Society of Cardiology recommendations alone
  n=46

INTERVENTIONS:
Behavioral: DISCO Intervention — optimal medical management in accordance with European Society of Cardiology recommendations + dietary intervention based on Dietary Approaches to Stop Hypertension (DASH diet) + strict monitoring of eating and lifestyle behaviors
  Groups: DISCO Intervention

SUMMARY:
A long-term evaluation of the impact of intensive diet and lifestyle intervention on coronary plaque dynamics in patients with coronary atherosclerosis diagnosed in computed tomography angiography (CCTA).

92 patients who completed the Dietary Intervention to Stop COronary Atherosclerosis in Computed Tomography study (DISCO-CT, NCT02571803) will be followed-up.

DETAILED DESCRIPTION:
All patients who completed the Dietary Intervention to Stop COronary Atherosclerosis in Computed Tomography received dietary and lifestyle recommendations and were referred to outpatient specialist care at their place of residence.

As part of this study, patients will be invited for a follow-up visit consisting of a cardiological and dietician consultation and additional tests, including CCTA, to assess the long-term impact of the intervention on the progression of atherosclerotic plaques, including high-risk plaque component.

Additionally, the occurrence of cardiovascular events, change in laboratory parameters and change in body weight composition will be analyzed.

ELIGIBILITY:
Inclusion criteria:

* completion the DISCO-CT study (NCT02571803)
* willingness to participate in the long-term follow-up at site

Exclusion criteria:

* contraindications to perform coronary computed tomography angiography (history of severe reaction to iodine contrast media, uncontrolled thyreotoxicosis and/or severe renal impairment with glomerular filtration rate < 30 ml/min)
* no consent to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be a group of participants of the DISCO-CT study (NCT02571803) who will be willing to participate in the long-term follow-up at site.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-01-13 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Total Atheroma Volume (Change) | 60 months
  Quantitative assessment of the coronary plaque dynamics will be analyzed in the coronary computed tomography angiography and compared with parameters measured at the completion of the DISCO-CT study (expressed in mm3)
Percent Atheroma Volume (PAV) (Change) | 60 months
  Quantitative assessment of the coronary plaque dynamics will be analyzed in the coronary computed tomography angiography and compared with parameters measured at the completion of the DISCO-CT study (expressed in percent)
  PAV = [(EEM-LA)/EEM]*100%
  EEM - external elastic membrane area LA - lumen area

SECONDARY OUTCOMES:
Calcified Plaque Volume (Change) | 60 months
  Analyzed in the coronary computed tomography angiography and compared with parameters measured at the completion of the DISCO-CT study; calcified plaque volume (expressed in mm3) will be identified according to plaque density in Hounsfield units, on a per-patient basis
Fibrous Plaque Volume (Change) | 60 months
  Analyzed in the coronary computed tomography angiography and compared with parameters measured at the completion of the DISCO-CT study; fibrous plaque volume (expressed in mm3) will be identified according to plaque density in Hounsfield units, on a per-patient basis
Fibrofatty Plaque Volume (Change) | 60 months
  Analyzed in the coronary computed tomography angiography and compared with parameters measured at the completion of the DISCO-CT study; fibrofatty plaque volume (expressed in mm3) will be identified according to plaque density in Hounsfield units, on a per-patient basis
Necrotic Core (Low Density) Plaque Volume (Change) | 60 months
  Analyzed in the coronary computed tomography angiography and compared with parameters measured at the completion of the DISCO-CT study; necrotic (low density) plaque volume (expressed in mm3) will be identified according to plaque density in Hounsfield units, on a per-patient basis
Non-Calcified Plaque Volume (Change) | 60 months
  Analyzed in the coronary computed tomography angiography and compared with parameters measured at the completion of the DISCO-CT study;
  A combined component of fibrofatty + necrotic (low density) plaque (expressed in mm3), measured on a per-patient basis
Rate of major cardiovascular events | 60 months
  * myocardial infarction
  * cardiovascular death
  * coronary revascularization

OTHER OUTCOMES:
Change in body mass | 60 months
  in kilograms
Change in total body fat | 60 months
  expressed in kilograms
Change in skeletal muscle mass | 60 months
  expressed in kilograms
Change in fat to muscle ratio | 60 months
  expressed as the relation of fat mass to muscle mass
Change in epicardial fat volume | 60 months
  semiautomated measurements based on the density in Hounsfield units performed in computed tomography angiography and expressed in cm3
Change in Visceral Fat Area | 60 months
  Measured as part of body composition analysis, expressed in cm2
Change in total cholesterol | 60 months
  mg/dL
Change in low density lipoprotein | 60 months
  mg/dL
Change in the DASH Index | 60 months
  adherence to the DASH plan in 8 main groups of foodstuffs (cereal products, vegetables, fruits, dairy products, meat, nuts/seeds, fats/oils, and sweets), with a maximum score of 10 per group (total 0 to 80)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Henzel, Principal Investigator — National Institute of Cardiology
Locations (1):
- National Institute of Cardiology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henzel J, Kepka C, Kruk M, Makarewicz-Wujec M, Wardziak L, Trochimiuk P, Dzielinska Z, Demkow M. High-Risk Coronary Plaque Regression After Intensive Lifestyle Intervention in Nonobstructive Coronary Disease: A Randomized Study. JACC Cardiovasc Imaging. 2021 Jun;14(6):1192-1202. doi: 10.1016/j.jcmg.2020.10.019. Epub 2020 Dec 16. PMID 33341413